CLINICAL TRIAL: NCT01471340
Title: A 26-Week Randomized, Double-Blinded, Active Controlled Study Comparing the Safety of Mometasone Furoate/Formoterol Fumarate MDI Fixed Dose Combination Versus Mometasone Furoate MDI Monotherapy in Adolescents and Adults With Persistent Asthma (Protocol No. P06241 Also Known as P202)
Brief Title: A Serious Asthma Outcome Study With Mometasone Furoate/Formoterol Versus Mometasone Furoate in Asthmatics 12 Years and Over (P06241)
Acronym: SPIRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P06241; 2011-002142-13 (EudraCT Number); MK-0887A-202 (Other: Merck Protocol Number)
Record Dates: First submitted 2011-11-10; First posted 2011-11-16 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; Mometasone Furoate, Formoterol Fumarate Drug Combination; Albuterol; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mometasone Furoate/Formoterol MDI BID (Experimental): MF/F MDI BID (pooled MF/F MDI 200/10 mcg BID and MF/F MDI 400/10 mcg BID treatments)
  Interventions: Drug: Mometasone Furoate/Formoterol MDI 100/5 mcg; Drug: Mometasone Furoate/Formoterol MDI 200/5 mcg; Drug: Albuterol 90 mcg /salbutamol 100 mcg HFA MDI; Drug: Prednisone/prednisolone
- Mometasone Furoate MDI BID (Active Comparator): MF MDI BID (pooled from MF MDI 200 mcg BID and MF MDI 400 mcg BID treatments)
  Interventions: Drug: Mometasone Furoate MDI 100 mcg; Drug: Mometasone Furoate MDI 200 mcg; Drug: Albuterol 90 mcg /salbutamol 100 mcg HFA MDI; Drug: Prednisone/prednisolone

INTERVENTIONS:
Drug: Mometasone Furoate/Formoterol MDI 100/5 mcg — two inhalations BID
  Other Names: MK-0887A; Dulera/Zenhale
  Arms: Mometasone Furoate/Formoterol MDI BID
Drug: Mometasone Furoate/Formoterol MDI 200/5 mcg — two inhalations BID
  Other Names: MK-0887A; Dulera/Zenhale
  Arms: Mometasone Furoate/Formoterol MDI BID
Drug: Mometasone Furoate MDI 100 mcg — two inhalations BID
  Other Names: Asmanex
  Arms: Mometasone Furoate MDI BID
Drug: Mometasone Furoate MDI 200 mcg — two inhalations BID
  Other Names: Asmanex
  Arms: Mometasone Furoate MDI BID
Drug: Albuterol 90 mcg /salbutamol 100 mcg HFA MDI — use as needed for asthma symptoms
Drug: Prednisone/prednisolone — Oral prednisone/prednisolone used only as an emergency rescue medication at the discretion of the investigator

SUMMARY:
The purpose of this study is to test the safety of DULERA. DULERA is a pressurized metered-dose inhaler (MDI) that contains two drugs combined, namely mometasone and formoterol in a single inhaler. Mometasone is an inhaled corticosteroid (ICS), which reduces the inflammation in the airways. Formoterol is a long-acting beta 2 agonist (LABA), which helps to relax the muscles of the airways in the lungs, making it easier to breathe. In combination, mometasone and formoterol are used for the treatment of asthma. This study will evaluate whether participants taking a LABA in combination with an ICS in a single inhaler have a different risk of having serious asthma events (hospitalization, intubation and death) compared to participants taking an ICS alone. The primary safety hypothesis is that the time-to-first serious asthma outcome (SAO) with mometasone furoate/formoterol (MF/F) MDI twice daily (BID) is non-inferior to that with mometasone furoate (MF) MDI BID in adolescents and adults with persistent asthma. If non-inferiority is achieved, the key secondary safety hypothesis of superiority of MF/F over MF will be assessed.

DETAILED DESCRIPTION:
Amendments 2 and 3 are specific to Brazil; all other countries will enroll patients under Amendment 1.

ELIGIBILITY:
Inclusion Criteria:

* Persistent asthma for at least 1-year
* Must use a daily asthma controller medication for at least 4 weeks prior to randomization, including an inhaled corticosteroid (ICS) with or without a long-acting beta agonist (LABA) or other adjunctive asthma therapy OR be using a leukotriene receptor antagonist (LTRA), xanthine or short acting beta agonist (SABA) as a monotherapy.
* Must be able to discontinue current asthma medication
* Must have a history of at least one asthma exacerbation in previous 4 to 52 weeks

Exclusion Criteria:

* Unstable asthma
* Taking high dose ICS with or without other adjunctive therapy who have an Asthma Control Questionnaire 6 (ACQ6) total score ≥ 1.5
* Taking LTRA, xanthine or SABA monotherapy with an ACQ-6 total score < 1.5 (controlled)
* Chronic obstructive pulmonary disease (COPD), cystic fibrosis (CF), or other significant, non-asthmatic, lung disease
* Clinically significant abnormality, illness or disorder of any body or organ system
* Significant underlying cardiovascular condition which may contraindicate use of a beta-agonist.
* History of smoking greater than 10-pack years
* Had an asthma exacerbation within 4 weeks of the Baseline Visit
* Had more than 4 asthma exacerbations or 2 hospitalizations within 52 weeks of the randomization visit
* Known or suspected hypersensitivity or intolerance to corticosteroids, beta-2 agonists, or any of the (inactive ingredients) excipients present in the medications used in this study
* Require the use of chronic systemic steroids, omalizumab, or other monoclonal or polyclonal antibodies
* Requires the use of beta-blockers
* History of life-threatening asthma, including an asthma episode that required intubation and/or was associated with hypercapnia requiring noninvasive ventilatory support
* Lactating, pregnant, or plans to become pregnant during the course of the trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11744 (Actual)
Dates: Start 2012-01-09 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weinstein CLJ, Ryan N, Shekar T, Gates D, Lane SJ, Agache I, Nathan RA; SPIRO Investigators. Serious asthma events with mometasone furoate plus formoterol compared with mometasone furoate. J Allergy Clin Immunol. 2019 Apr;143(4):1395-1402. doi: 10.1016/j.jaci.2018.10.065. Epub 2018 Dec 8. PMID 30537475
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11,744 participants were enrolled in the study and 11,729 participants were randomized and received at least one dose of blinded study treatment (defined as the number started). Treatments were Mometasone Furoate/Formoterol (MF/F) metered dose inhaler (MDI) twice daily (BID) and Mometasone Furoate (MF) MDI BID.
Groups:
- Mometasone Furoate/Formoterol (MF/F) MDI BID: MF/F MDI administered as two puffs of 100/5 mcg or 200/5 mcg, twice daily (pooled MF/F treatments), with oral inhalation of a pressurized inhalation aerosol
- Mometasone Furoate (MF) MDI BID: MF MDI administered as two puffs of 100 mcg or 200 mcg, twice daily (pooled MF treatments), with oral inhalation of a pressurized inhalation aerosol
Period: Overall Study
Arm/Group | Mometasone Furoate/Formoterol (MF/F) MDI BID | Mometasone Furoate (MF) MDI BID
Started | 5868 (This value corresponds to randomized participants who received at least of dose of study medication) | 5861 (This value corresponds to randomized participants who received at least of dose of study medication)
Completed | 5862 | 5855
Not Completed | 6 | 6
Not completed — Death | 5 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Investigational site closure | 0 | 1
Not completed — Invalid informed consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: These are all participants who were randomized and treated with at least one dose of study medication
Groups:
- Mometasone Furoate/Formoterol (MF/F) MDI BID: MF/F MDI administered as two puffs of 100/5 mcg or 200/5 mcg, twice daily, with oral inhalation of a pressurized inhalation aerosol
- Mometasone Furoate (MF) MDI BID: MF MDI administered as two puffs of 100 mcg or 200 mcg, twice daily, with oral inhalation of a pressurized inhalation aerosol
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate/Formoterol (MF/F) MDI BID | Mometasone Furoate (MF) MDI BID | Total
Number analyzed (Participants) | 5868 | 5861 | 11729
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.3 (17.19) | 44.8 (17.55) | 45.1 (17.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3841 | 3875 | 7716
  Male | 2027 | 1986 | 4013
Treatment Covariates (MF/F or MF) and ICS Dose Level (100 or 200 mcg, per actuation) [Count of Participants; unit: Participants] — The primary safety hypothesis will be evaluated using Cox proportional-hazard model including covariates of treatment (MF/F MDI BID vs MF MDI BID) and ICS dose level (100 mcg vs 200 mcg, per actuation).
  Participants
    MF/F 200/10 mcg | 3604 | 0 | 3604
    MF/F 400/10 mcg | 2264 | 0 | 2264
    MF 200 mcg | 0 | 3601 | 3601
    MF 400 mcg | 0 | 2260 | 2260

OUTCOME MEASURES:

1. Primary Outcome: Time-to-First Serious Asthma Outcomes (SAO): Number of First SAO in the MF/F vs MF Arms
Description: The primary safety outcome was the time-to-first SAO (a composite endpoint of adjudicated asthma-related hospitalizations, adjudicated asthma-related intubations, and adjudicated asthma-related deaths). To accomplish this, the number of participants experiencing a first SAO was collected for 26 weeks following initiation of study treatment (or 7 days after the last treatment dose, whichever occurred later). Data generated by this methodology were used to compute a hazard ratio (HR) and 95% confidence interval (CI), modeling the likelihood of a first SAO occurring at any given time in the MF/F arm relative to the MF arm. Although data were sufficient to generate a HR and 95% CI, time-to-first SAO in the overall population could not be accurately reported due to insufficient SAO occurrence. Therefore, the number of first SAO in either arm is reported as a descriptive measure. For each participant, first SAO denotes first event per participant.
Time Frame: 26 weeks, or 7 days after the last treatment dose, whichever occurred later
Population: The analyzed population for assessment of the number of first SAO was all participants who received at least one dose of randomized treatment assignment (intention-to-treat principle).
Measure: Number; unit: Serious asthma outcomes
Groups:
- MF/F MDI BID: MF/F MDI administered as two puffs of 100/5 mcg or 200/5 mcg, twice daily (pooled MF/F treatments), with oral inhalation of a pressurized inhalation aerosol
- MF MDI BID: MF MDI administered as two puffs of 100 mcg or 200 mcg, twice daily (pooled MF treatments), with oral inhalation of a pressurized inhalation aerosol
Arm/Group | MF/F MDI BID | MF MDI BID
Number analyzed (Participants) | 5868 | 5861
Serious asthma outcomes | 39 | 32
Statistical Analysis 1: Comparison: MF/F MDI BID vs MF MDI BID; Pertains only to the First SAO; pooled MF/F treatments and pooled MF treatments; Test type: Non-Inferiority or Equivalence — The projected sample size provided 90% power at a 2.5% alpha level (one-sided) to determine non-inferiority of MF/F and MF. For analysis of the first SAO in participants, MF/F MDI BID was considered non-inferior to MF MDI BID if the upper bound for the 95% confidence interval (CI) of the hazard ratio (HR) of MF/F MDI BID versus MF MDI BID was lower than 2.0 (noninferiority margin); p = 0.411, Cox proportional-hazard model; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.76 to 1.94] — The HR and 95% CI were based on the Cox proportional-hazard model with covariates of treatment (MF/F or MF) and ICS dose level (200 or 400 mcg)

2. Secondary Outcome: Time-to-First Severe Asthma Exacerbation (SAEX): Number of First SAEX in the MF/F vs MF Arms
Description: The key secondary efficacy outcome was time-to-first protocol-defined asthma exacerbation (SAEX). The SAEX were deteriorations of asthma requiring: use of systemic corticosteroids (tablets, suspension, or injection) for >= 3 consecutive days, in-patient hospitalization >= 24 hours, or an emergency department (ED) visit < 24 hours that required systemic corticosteroids in the MF/F MDI BID arm versus the MF MDI BID arm. The number of first SAEX occurred from initiation of study treatment to 7 days after the last treatment (modified intention-to-treat). This outcome was measured as the HR and 95% CI for the number of first SAEX in the MF/F MDI BID arm versus the number of first SAEX in the MF MDI BID arm. Given insufficient data for SAEX events, it was not informative to report the time-to-first SAEX in the overall population. Therefore, the number of first SAEXs in either arm is reported as a descriptive measure. For each participant, first SAEX denotes first event per participant.
Time Frame: 26 weeks, plus 7 days after the last treatment
Population: The analyzed population for assessment of the number of first asthma exacerbations was all treated participants who received at least one dose of randomized treatment assignment (intention-to-treat principle).
Measure: Number; unit: Asthma exacerbations
Arm/Group | MF/F MDI BID | MF MDI BID
Number analyzed (Participants) | 5868 | 5861
Asthma exacerbations | 708 | 779
Statistical Analysis 1: Comparison: MF/F MDI BID vs MF MDI BID; Pertains only to the First SAEX; pooled MF/F treatments and pooled MF treatments; Test type: Superiority or Other; p = 0.021, Cox proportional-hazard model; Superiority of MF/F MDI BID vs MF MDI BID was determined if the HR was less than 1 and achieved statistical significance (one-sided p-value < 0.025); Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.80 to 0.98] — [estimate comment as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Number of SAO Components in MF/F Participants vs MF Participants
Description: To further examine the primary safety outcome, each adjudicated component of the SAO composite endpoint (asthma-related hospitalization, asthma-related intubation and asthma-related death), was tabulated for descriptive purposes only to show the relative contribution of each component to the SAO composite. Hospitalizations were defined as an in-patient stay of >= 24 hour in a hospital, emergency department or equivalent healthcare facility. Intubation was defined as endotracheal intubation only.
Time Frame: 26 weeks, or 7 days after the last treatment dose, whichever occurred later
Population: The analyzed population for tabulation of the number of SAO components was all participants who received at least one dose of randomized treatment assignment (intention-to-treat principle).
Measure: Number; unit: SAO components
Arm/Group | MF/F MDI BID | MF MDI BID
Number analyzed (Participants) | 5868 | 5861
SAO components
  First SAO | 39 | 32
  Asthma-related hospitalizations | 39 | 32
  Asthma-related intubations | 0 | 0
  Asthma-related deaths | 0 | 0

ADVERSE EVENTS:
Time Frame: 26 weeks, or 7 days after the last treatment dose, whichever occurred later
Description: All serious adverse events are reported. Only those non-serious (Other) adverse events leading to treatment discontinuation were collected during the study, and are reported here.
Arm/Group | MF/F MDI BID | MF MDI BID
All-Cause Mortality (participants affected / at risk) | 5/5868 | 4/5861
Serious Adverse Events (participants affected / at risk) | 136/5868 | 137/5861
Other Adverse Events (participants affected / at risk) | 67/5868 | 75/5861
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F MDI BID (N=5868) | MF MDI BID (N=5861)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric dysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1)
Anicteric leptospirosis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 6 (6) | 4 (4)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3) | 0 (0)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 2 (2) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 10 (11) | 6 (6)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional product misuse (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest X-ray abnormal (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperosmolar state (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Carcinoid tumour of the duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophreniform disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 32 (34) | 31 (34)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F MDI BID (N=5868) | MF MDI BID (N=5861)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 3 (3)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Feeling jittery (General disorders) | 1 (1) | 1 (1)
Tongue discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Laryngeal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchospasm paradoxical (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Hypopnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 7 (7)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Oral mucosal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Allergic edema (Immune system disorders) | 0 (0) | 1 (1)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor, and to provide the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication which report any trial results. The sponsor has the right to review and comment on publications, abstracts, slides, and manuscripts, and to review and comment on data analysis and presentation.